CLINICAL TRIAL: NCT00873262
Title: A Phase II Randomized, Two-arms, Single-blind, Cross Controlled Study for Evaluation the Safety and Efficacy of Diagnosis and Treatment of Premenstrual Syndrome by Detecting Skin Reactions Followed by Desensitization to Sex Hormones
Brief Title: Evaluation of Safety/Efficacy of Diagnostic Skin Test Panel and Desensitization Hormone Kit for Treatment of Premenstrual Syndrome (PMS)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: EVE Medical Systems Ltd. (Industry)
Responsible Party: Dr. Yonit Bomstein, EVE Medical Systems Ltd.
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: EVE-2008-03
Record Dates: First submitted 2009-03-30; First posted 2009-04-01 (Estimated); Last update posted 2010-06-16 (Estimated); Status verified 2010-02

CONDITIONS: Premenstrual Syndrome
Keywords: PreMenstrual Syndrome; Hormones; Skin tests; Desensitization; Allergen Immunotherapy
MeSH Terms: conditions — Premenstrual Syndrome | interventions — Progesterone; Estradiol; Estrone; Estriol; Solvents

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hormones (Active Comparator)
  Interventions: Drug: Skin test panel and desensitization kit
- Solvent (Placebo Comparator)
  Interventions: Drug: Skin test panel and solvent

INTERVENTIONS:
Drug: Skin test panel and desensitization kit — Skin testing 4 sex hormones will be performed during the luteal phase of the subject's menstrual cycle by study investigators.
  Hormones:
  Progesterone 1mmol/L; Estradiol 1mmol/L; Estrone 3mmol/L; Estriol 3mmol/L
  Controls:
  Saline (NaCl) 0.9%; Ethyl Oleate with 10% Benzyl Alcohol; Histamine phosphate 1mg/ml (epicutaneous- prick test)
  Patients with positive skin test to at least one sex hormone will be injected with an increasing volume of the appropriate hormone at the same concentration as it was used in the skin test as follows:
  1. Week 4th of the study (luteal phase of 2nd menstrual cycle) - 0.04 ml
  2. Week 8th of the study (luteal phase of 3rd menstrual cycle) - 0.08 ml
  3. Week 12th of the study (luteal phase of 4th menstrual cycle) - 0.16 ml
  Other Names: Progesterone; Estradiol; Estrone; Estriol
  Arms: Hormones
Drug: Skin test panel and solvent — Skin testing 4 sex hormones will be performed during the luteal phase of the subject's menstrual cycle by study investigators.
  Hormones:
  Progesterone 1mmol/L; Estradiol 1mmol/L; Estrone 3mmol/L; Estriol 3mmol/L
  Controls:
  Saline (NaCl) 0.9%; Ethyl Oleate with 10% Benzyl Alcohol; Histamine phosphate 1mg/ml (epicutaneous- prick test)
  Patients with positive skin test to at least one sex hormone will be injected with an increasing volume of the solvent as follows:
  1. Week 4th of the study (luteal phase of 2nd menstrual cycle) - 0.04 ml
  2. Week 8th of the study (luteal phase of 3rd menstrual cycle) - 0.08 ml
  3. Week 12th of the study (luteal phase of 4th menstrual cycle) - 0.16 ml
  Other Names: Progesterone; Estradiol; Estrone; Estriol
  Arms: Solvent

SUMMARY:
The EVE-PMS technology is intended for determination of intolerance or sensitivity to sex hormones, among women suffering from severe PreMenstrual Syndrome (PMS) and desensitizes them with the relevant sex hormones in order to reduce PMS symptoms.

The system includes skin testing panel for identification of hormones to which the patients might be sensitive. Tests are applied close to the ovulation period and the skin reaction is examined in 20 minutes, 48 hours and daily during the following month. Results of skin tests and patient's history will determine the eligibility of the patients to enter a desensitization protocol.

During the desensitization period hormones to which the patient were found sensitive to, are injected intradermally three times (once a month) within the luteal phase in increasing doses. The end-point of the study is a statistically significant decrease, or elimination of PMS symptoms, compared to a solvent group.

ELIGIBILITY:
Inclusion Criteria:

1. Person is over the age of 20 but not older than age 45.
2. Person is willing to participate as evidenced by signing the written informed consent form.
3. Suffers from known dominant severe symptom of breast swelling and tenderness (level 7-10 according to standard scale of PMS symptoms severity)
4. Other severe symptoms of Premenstrual syndrome (based on WHO and ACOG criteria). This may include one or more of PMS symptoms with level 7-10 according to standard scale of PMS symptoms severity.
5. At work, school, home, or in daily routine, at least one of the PMS symptoms caused reduction of productivity or inefficiency
6. At least one of the PMS symptoms caused avoidance of or less participation in hobbies or social activities
7. At least one of the PMS symptoms interfere with relationships with others

   * Timing of PMS symptom(s): during the 14 days prior to onset of menstrual flow (rather than spotting) and up to 5 days during the menstrual flow.
   * Pattern and length of PMS symptomatic period: minimum of 2 days, up to 14 days.
   * For PMS diagnosis two out of last three consecutive menstrual cycles were monitored by daily monitoring of symptoms.
   * Timing and length of asymptomatic phase: day 6 to at least day 10 of the menstrual cycle.
   * Cyclicity - presentation of the 'off-on' phenomenon: there should be a clear shift from no PMS symptoms to PMS symptoms.
   * Reliable non hormonal contraception.

Exclusion Criteria:

1. Pregnant or lactating woman
2. Oral contraceptives during last three months, including hormonal IUD (trade name mirena).
3. Serious health problems.
4. Unexplained menstrual disorders.
5. Treated by hormones (estrogen and progesterone).

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2009-04; Primary Completion 2010-05 (Estimated); Study Completion 2010-11 (Estimated)

PRIMARY OUTCOMES:
To assess the efficacy of hormonal desensitization compared to solvent treatment in reduction of the PMS symptoms severity and length of PMS by subjects with severe PMS symptoms (according to criteria of PMS). | 5-6 months

SECONDARY OUTCOMES:
To assess the efficacy of hormonal desensitization compared to solvent treatment in reduction of the breast swelling and tenderness in 4 weeks of treatment. | 2-3 months

CONTACTS AND LOCATIONS:
Overall Officials: Shmuel Kivity, Prof., Principal Investigator — Tel Aviv Sourasky Medical Center, Department of Allergy and clinical immunology; Jacob Cohen, Dr., Principal Investigator — Tel Aviv Sourasky Medical Center, Department of Outpatient Gynecology Clinics
Locations (1):
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel